CLINICAL TRIAL: NCT06515314
Title: A Phase 1, Single-arm, Open-label, Dose-escalation Study of AFP Specific T Cell Receptor Transduced T Cells Injection（HRYZ-T102）in Patients With AFP Positive Advanced Hepatocellular Carcinoma and Other Solid Tumors
Brief Title: HRYZ-T102 TCR-T Cell for AFP Positive Advanced HCC and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ruiliyuan Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-T02-C1001
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRYZ-T102 Injection (Experimental): Patients will undergo lymphocytapheresis, then treatment with HRYZ-T102 TCR-T cells.
  Interventions: Biological: AFP Specific T Cell Receptor T Cells

INTERVENTIONS:
Biological: AFP Specific T Cell Receptor T Cells — AFP Specific T Cell Receptor T Cells On day 1, the TCR-T cells will be administered intravenously.
  Drug: Fludarabine + Cyclophosphamide Fludarabine: 25mg/m²/day×3days; Cyclophosphamide: 250mg/m²/day×3 days

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and efficacy of HRYZ-T102 TCR-T Cell in patients with AFP positive advanced hepatocellular carcinoma and other solid tumors refractory to prior systematic treatments.

DETAILED DESCRIPTION:
This study plans to enroll 12-24 patients to assess the safety of HRYZ-T102. Subjects who meet the eligibility criteria will receive a single dose of HRYZ-T102 injection .The patient will be followed up 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be willing to sign the informed consent form.
2. Age ≥18 years and ≤75 years.
3. HLA-A 02:03 allele positive
4. Histologically-confirmed AFP positive hepatocellular carcinoma (HCC) or other solid tumor, No benefits from curative surgery or other local therapies are expected ,at least one prior line of systematic treatment at screening, judged by investigators.
5. Fresh samples or formalin-fixed paraffin-embedded (FFPE) samples, immunohistochemistry (IHC)-stained AFP positive or serum AFP ≥400ng/ml.
6. Barcelona Clinic Liver Cancer (BCLC) stage C or B and Child-Pugh ≤7
7. ECOG performance status ≤1.
8. Estimated life expectancy ≥4 months.
9. Patients must have at least one measurable lesion defined by RECIST 1.1.
10. Patients with any organ dysfunction as defined below:

    Leukocytes≥3.0 x 10^9/L; blood platelets ≥75 x 10^9/L; hemoglobin≥85g/L; Absolute lymphocyte count≥0.8 x 10^9/L Serum albumin ≥ 30g/L; total bilirubin≤3×ULN; ALT/AST≤3×ULN ; Creatinine clearance ≥50mL/min; or serum creatinine ≤1.5×ULN; INR≤1.5×ULN; APTT≤1.5×ULN; LVEF≥50%; SpO2≥92%.
11. Subjects with potential fertility must agree to use effective contraceptive methods during the whole trials period and at least 1 year after receiving HRYZ-T102 cell transfusion treatment. HCG test for female with potential fertility must be negative within 7 days before apheresis.

Exclusion Criteria:

1. Toxicity of previous treatment has not been mitigated or ≤ Grade 1 at screening.
2. Another primary malignancy within 5 years (with some exceptions for completely-resected early-stage tumors)
3. With severe cardiovascular disease or presence of clinically-relevant central nervous system (CNS) disorders in six months before screening.
4. Systematic autoimmune disorders requiring long-term systematic immunosuppression
5. Have a history of hypersensitivity to cyclophosphamide or fludarabine, and it is known that any ingredient used in the treatment of this study will produce allergic reactions.
6. Current presence of or previously with hepatic encephalopathy
7. Organ transplanters and allogeneic cell transplanters.
8. Have a history of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within 3 months before screening
9. Hereditary or acquired bleeding (e.g. coagulation dysfunction) or a tendency to clot
10. Subject has active infection or unexplained fever during screening and prior to cell transfusion
11. Have central nervous system metastasis with symptoms
12. Known HIV or syphilis infection, and/or active hepatitis C virus infection.
13. HBV infect subjects with HBV-DNA≥2000IU/ml
14. Pregnant or lactating female, or those whose HCG test is positive before enrollment.
15. Known uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | 2 years
  Incidence of adverse events and serious adverse events
DLT | 2 years
  Dose-limiting toxicity

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  The percentage of subjects with PR or CR assessed by RECIST 1.1.
Disease Control Rate (DCR) | 2 years
  The percentage of subjects with a confirmed CR, PR, or stable disease (SD) assessed by RECIST 1.1.
Duration of response (DoR) | 2 years
  Subjects who show a confirmed CR or PR as assessed by RECIST 1.1.
Time to response (TTR) | 2 years
  Time from date of T-cell administration to first documented evidence of confirmed (CR or PR) as assessed by RECIST 1.1.
Progression-Free Survival（PFS） | 2 years
  The length of time from enrollment until the time of progression of disease
Overall Survival (OS) | 2 years
  The interval of time between the date of T-cell infusion and the date of death.
Duration of TCR T cells in-vivo persistence | 2 years
  Blood samples were collected to measure persistence of infused HRYZ-T102
Concentration of Cytokines (IL-2、IL-6、IL-10、TNFα、IFNγ) | 2 years
  Collect blood samples and analyze for presence of cytokines (IL-2、IL-6、IL-10、TNFα、IFNγ) at specified intervals before and after treatment with HRYZ-T102.

OTHER OUTCOMES:
Number of Subjects with positive anti-drug antibodies (ADA) | 2 years
  Serum samples will be collected to analyze for the presence of ADAs using validated immunoassays
Number of subjects with replication competent lentivirus (RCL) | 2 years
  RCL exposure will be assessed by polymerase chain reaction (PCR) based assay.
T cell subgroup in peripheral blood | 2 years
  Collect blood samples and analyze for T cell subgroup by flow cytometry at specified intervals before and after treatment with HRYZ-T102.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowu Huang, Doctor, Principal Investigator — Study Principal Investigator
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China